CLINICAL TRIAL: NCT04714229
Title: A Single Center, Randomized, Observer-blinded, Active Comparator Phase I Study to Assess the Safety and Immunogenicity of Meningococcal (Groups A, C, W-135 and Y) Conjugate Vaccine in Healthy Adults Aged 19 to 55 Years Old
Brief Title: Safety and Immunogenicity of Meningococcal Conjugate Vaccine in Healthy Adults Aged 19 to 55 Years Old
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: EuBiologics Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: EuVCT_MCV101
Record Dates: First submitted 2021-01-14; First posted 2021-01-19 (Actual); Last update posted 2021-10-07 (Actual); Status verified 2021-01

CONDITIONS: Infection, Meningococcal
MeSH Terms: conditions — Meningococcal Infections | interventions — Vaccines, Conjugate; Meningococcal Vaccines

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EuMCV4 (Experimental): Healthy adults received 0.5mL single intramuscular dose on Day 0.
  Interventions: Biological: Meningococcal(Groups A, C, W-135, and Y) Conjugate Vaccine
- Menveo (Active Comparator): Healthy adults received 0.5mL single intramuscular dose on Day 0.
  Interventions: Biological: Meningococcal(Groups A, C, Y, and W-135) Conjugate Vaccine

INTERVENTIONS:
Biological: Meningococcal(Groups A, C, W-135, and Y) Conjugate Vaccine — 0.5mL single intramuscular dose on Day 0
  Other Names: EuMCV4
  Arms: EuMCV4
Biological: Meningococcal(Groups A, C, Y, and W-135) Conjugate Vaccine — 0.5mL single intramuscular dose on Day 0
  Other Names: Menveo
  Arms: Menveo

SUMMARY:
Phase I study to evaluate safety and immunogenicity in healthy adult subjects following a single dose administration of Meningococcal (Group A, C, W-135, and Y)-CRM197 Conjugate vaccine

ELIGIBILITY:
Inclusion Criteria:

* Subjects 19 to 55 years of age
* Written informed consent
* Available for all visits and telephone calls scheduled for the study

Exclusion Criteria:

* Previous or suspected disease caused by N. meningitidis
* Household and/or intimate exposure to an individual with culture-proven N. meinigitidis infection within 60 days prior to screening
* Serious acute, chronic or progressive disease as determined by investigator
* History of alcohol or substance abuse

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2020-11-01 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
Occurrence of solicited adverse events | within 7 days post vaccination
  local and systemic AEs
Occurrence of unsolicited adverse events | within 28 days post vaccination
Occurrence of serious adverse events | within 180 days post vaccination

CONTACTS AND LOCATIONS:
Overall Officials: YJ Lee, Study Director — EuBiologics Co.,Ltd
Locations (1):
- Seoul National University Hospital, Seoul, South Korea